CLINICAL TRIAL: NCT05995015
Title: Universal 4SCAR19U T Cell Therapy for the Treatment of Relapsed and Refractory B Cell Malignancies
Brief Title: 4SCAR19U T Cells Targeting B Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-23001
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: B Cell Malignancies
Keywords: Universal CAR-T; CD19 B-ALL; PMBCL; CNS-BCL; BCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Universal 4SCAR19U cells to treat CD19-positive hematological malignancies (Experimental)
  Interventions: Biological: Universal CD19-specific CAR gene-engineered T cells

INTERVENTIONS:
Biological: Universal CD19-specific CAR gene-engineered T cells — Infusion of 4SCAR19U cells

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of universal CAR T cell therapy against CD19-positive hematological malignancies using a novel CD19-specific CAR T cell product, 4SCAR19U T cells. The study also aims to learn more about the function of the 4SCAR19U T cells and their persistence in patients. This is a phase I trial enrolling patients from multiple clinical centers.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cell therapy has proven effective in treating B cell malignancies. However, the application itself is still limited by the high cost and long preparation time which often do not meet the urgent need of patients. In addition, some patients may suffer from long-term immunosuppression caused by tumor microenvironment or after radiotherapy and chemotherapy, resulting in exhaustion, aging and functional defects of the autologous T cells, which will eventually affect the quality of the CAR-T cells and affect the clinical efficacy.

The 4SCAR19U T cells are genetically engineered and manufactured in bulk amount that can be supplied off-the-shelf without being custom made from individual patients. The immediate availability of the CAR-T cells makes clinical treatment convenient and timely for rapid progressing disease or for the highly immune suppressed patients. This application can be time- and cost-effective. This novel approach may also overcome problems of functionally defective autologous T cells. The purpose of this clinical trial is to assess the feasibility, safety and efficacy of the 4SCAR19U T cell product in hematological malignancies. Another goal of the study is to learn more about the function of this novel product and its persistence in the patients

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Primary B cell surface expression of CD19.
3. The KPS score over 80 points, and survival time is more than 1 month.
4. Greater than Hgb 80 g/L.
5. No contraindications to blood cell collection.

Exclusion Criteria:

1. Accompanied with other active diseases, and difficult to assess response after treatment.
2. Bacterial, fungal, or viral infection, unable to control.
3. Living with HIV.
4. Active HBV or HCV infection.
5. Pregnant and nursing mothers.
6. under systemic steroid treatment within a week of the treatment.
7. Prior failed CAR-T treatment.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of 4SCAR19U CAR-T cells infusion | 24 weeks
  Safety of 4SCAR19U T cells in patients with relapsed and refractory B-ALL, BCL using CTCAE 4 standard to evaluate the level of adverse events

SECONDARY OUTCOMES:
Anti-tumor activity of 4SCAR19U cells after infusion | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No